CLINICAL TRIAL: NCT04082403
Title: The Impact of Suction- Assisted Laryngoscopy and Airway Decontamination on Intubation Times
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dylan Finnerty (Other)
Responsible Party: Sponsor-Investigator, Dylan Finnerty, Anesthesia Specialist Registrar, Mater Misericordiae University Hospital
Organization: Mater Misericordiae University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MaterMUH2019
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Contaminated Airway

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre SALAD education group (Active Comparator): Each trainee was asked to intubate a mannequin with a contaminated airway
  Interventions: Procedure: No Training on Suction Assisted Laryngoscopy and Airway Decontamination Provided
- Post SALAD education group (Experimental): Each trainee was asked to intubate a mannequin with a contaminated airway after receiving SALAD training
  Interventions: Procedure: Training on Suction Assisted Laryngoscopy and Airway Decontamination

INTERVENTIONS:
Procedure: Training on Suction Assisted Laryngoscopy and Airway Decontamination — Education on Suction Assisted Laryngoscopy and Airway Decontamination, via 30 minute teaching session, followed by practical demonstration of techniques.
  Arms: Post SALAD education group
Procedure: No Training on Suction Assisted Laryngoscopy and Airway Decontamination Provided — No Training on Suction Assisted Laryngoscopy and Airway Decontamination provided to trainees
  Arms: Pre SALAD education group

SUMMARY:
A study was formulated to test the hypothesis that comprehensive training in Suction- Assisted Laryngoscopy and Airway Decontamination techniques reduces mannequin intubation times for Anaesthesia trainees.

DETAILED DESCRIPTION:
To assess the clinical impact of in Suction- Assisted Laryngoscopy and Airway Decontamination (SALAD) training among 37 anaesthesia trainees. Intubation mannequin will be used to assess intubation times for contaminated airways pre and post SALAD training.

ELIGIBILITY:
Inclusion Criteria:

All Anaesthesia trainees employment in Mater Misericordiae University hospital during the month of August 2019 - October 2019 were invited to partake in the study.

Exclusion Criteria:

All intensive care trainees with no training in intubation were excluded from the study.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2019-09-19 (Estimated); Primary Completion 2019-10-19 (Estimated); Study Completion 2019-10-19 (Estimated)

PRIMARY OUTCOMES:
Time to intubation as preformed on a mannequin . | 1 month
  Aim to investigate whether specific airway training on contaminated airways reduced intubation time in anaesthesia trainees.

IPD SHARING:
Plan to Share IPD: No